CLINICAL TRIAL: NCT03645044
Title: Towards a Functional Cure for HBV: Exploiting Lessons From HIV-HBV Co-infection: The COMMIT Cohort Study
Brief Title: Towards a Functional Cure for HBV - The COMMIT Cohort Study
Acronym: COMMIT
Status: Active, not recruiting | Type: Observational
Sponsor: University of Melbourne (Other)
Collaborators: National Health and Medical Research Council, Australia (Other); The University of Western Australia (Other); University of Adelaide (Other); The HIV Netherlands Australia Thailand Research Collaboration (Other); University of Malaya (Other); YR Gaitonde Centre for AIDS Research and Education (Other); Melbourne Health (Other)
Responsible Party: Principal Investigator, Joe Sasadeusz, Infectious Diseases physician, University of Melbourne
Other Study IDs: COMMIT study (NMHRC 1123988)
Record Dates: First submitted 2018-08-22; First posted 2018-08-24 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Hiv; HBV Coinfection
Keywords: HBV sAg loss/seroconversion; HBV "e" antigen (eAg) loss/seroconversion; antiretroviral therapy
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — peripheral blood mononuclear cells (PBMCs) and plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hepatitis B virus (HBV) infection can be treated, but therapy is usually lifelong and has side effects, so a cure for HBV is a critical endpoint. This study examines the key steps to HBV cure in the setting of HIV-HBV co-infection, where rates of development of antibodies against HBV after starting HBV treatment are higher than in people with HBV alone starting treatment. In Asia both HBV and HIV are common so this provides a unique opportunity to study HBV. We will investigate how an effective immune response against the two main HBV proteins is developed. If we can understand how the immune response works against HBV, this could be used to develop new therapies towards a cure for HBV

DETAILED DESCRIPTION:
A) Aims and Objectives. Effective antiviral treatments of HBV are available, but treatment is lifelong in most so comes at considerable cost and with some toxicity. An effective therapeutic strategy to achieve a cure for HBV remains an unmet need. This project examines the key steps to HBV cure in the setting of HIV-HBV co-infection. Seroconversion is key to the cure. Seroconversion is the process where detectable antibody (specific protective protein produced by the immune system) against virus proteins (antigens) are developed in the blood. This proposed Asian HIV-HBV co-infection cohort (where treatment initiation is later and hence at lower cluster of differentiation 4 (CD4) counts) will provide a unique opportunity to test our hypothesis that following initiation of antiviral therapy, HB surface and "e" antigen loss is more frequent (i) early in treatment and (ii) with lower CD4 cell counts, and that predictors of losing HB surface and 'e" antigen (Ag) and gaining antibody (Ab) against them are directly associated with B-cell functions.

B) Key Questions. Primary objective: to determine the rates & clinical determinants of HBsAg and HBeAg loss and seroconversion in HIV-HBV co-infected patients commencing HBV-active antiretroviral (ART). We will test the hypotheses that: (i) seroconversion occurs predominantly in the early phase of treatment (≤12 months) with HBV active ART and (ii) seroconversion is more frequent in HIV-HBV co-infected individuals commencing treatment with lower CD4+ T cell counts (≤100 cells/mm3) compared to those with higher counts (>100 cells/mm3).

Secondary objectives: (i) identify predictive biomarkers of HBsAg loss/seroconversion and (ii) examine predictors of HBeAg loss/seroconversion in this setting

C) Research Design. This is a large prospective, observational cohort study of treatment-naïve HIV-HBV co-infected patients (n=150). Clinical sites are - (1) HIV-Netherland-Australia-Thailand (HIV-NAT)/Thai Red Cross AIDS Research Centre, Bangkok, Thailand; (2) Y.R. Gaitonde Centre for AIDS Research and Education (YRG CARE), Chennai, India; and (3) Clinical Investigation Centre (CIC), University of Malaya, Infectious Diseases Directorate, Kuala Lumpur, Malaysia. Participants will be followed for 2 years, with study visits at baseline (study entry/initiation of treatment), months 3, 6, 12, 18, and 24 of follow-up. Clinical and laboratory information/data and blood samples will be collected at study visits.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 years and older
* HIV antibody positive
* Chronically-infected with HBV, as defined by:

  i. Positive Hepatitis B surface antigen HBsAg) or HBV DNA result with a subsequent positive HBsAg or HBV DNA result at least 6 months after first positive result (the 2nd HBsAg test may be taken at the baseline visit) ii. HBsAg positive with the absence of immunoglobulin M antibodies to HBV core at screening
* Current or ever hepatitis C virus (HCV) antibody negative
* Hepatitis D virus (HDV) negative
* ART naïve or within 7-10 days of ART start at sites where immediate ART start (test and treat) is practice
* Provide signed and dated informed consent form.
* Willing to comply with all study procedures and be available for the duration of the study.

Exclusion Criteria:

* Hepatitis C virus (HCV) antibody positive
* Hepatitis delta antibody positive
* Anything that would place the individual at increased risk or preclude the individual's full compliance with or completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Anti-retroviral treatment (ART) naïve (or within 7-10 days of ART start where immediate ART start (test and treat) is practice) HIV-HBV co-infected individuals about to commence ART, aged 18 years and older
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2018-05-24 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
HBsAg loss/seroconversion on ART | 24 months
  Frequency of HBsAg loss/seroconversion in early (first 12 months) compared to later stage

SECONDARY OUTCOMES:
HBeAg loss/seroconversion on ART | 24 months
  Frequency of HBeAg loss/seroconversion in early (first 12 months) compared to later stage
HBsAg epitope profiles | 24 months
  HBsAg epitope profiles at study entry and after 2 years of antiviral therapy in HBsAg responders and non-responders
Differential B cell gene expression | 24 months
  Differential B cell gene expression (genetic testing) in HBsAg responders and non-responders after 2 years of antiviral therapy
B-cell activating factor (BAFF) levels | 24 months
  Levels of BAFF in plasma at study entry and after 2 years of antiviral therapy in HBsAg responders and non-responders
HBeAg and HBsAg specific memory B cells | 24 months
  Proportion of HBeAg and HBsAg specific memory B cells at study entry and after 2 years of antiviral therapy
B cell subtypes | 24 months
  Percentage of B cell subtypes at study entry and after 2 years of antiviral therapy

CONTACTS AND LOCATIONS:
Overall Officials: Joe Sasadeusz, MBBS, PhD, Principal Investigator — University of Melbourne
Locations (3):
- YRGCare, Chennai, India
- Clinical Investigation Centre (CIC), University of Malaya, Infectious Diseases Directorate, Kuala Lumpur, Malaysia
- HIV-NAT/Thai Red Cross AIDS Research Centre, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No